CLINICAL TRIAL: NCT02854241
Title: Comparison of Biannual Ultrasonography and Annual Unenhanced Magnetic Resonance Imaging as a Surveillance Test for HCC in Patients With Liver Cirrhosis
Brief Title: Comparison of Biannual Ultrasonography and Annual Unenhanced Magnetic Resonance Imaging for HCC Surveillance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SNUH-2016-0174
Record Dates: First submitted 2016-07-31; First posted 2016-08-03 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cirrhosis; Hepatocellular Carcinoma
Keywords: MRI; HCC; surveillance
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LC group (Experimental): LC group under surveillance of biannual ultrasonography and annual noncontrast liver MRI. Six month after the last MRI, contrast enhanced liver CT is performed to investigate presence of HCC.
  Interventions: Procedure: Biannual ultrasonography; Procedure: Annual noncontrast liver MRI; Procedure: Contrast enhanced liver CT

INTERVENTIONS:
Procedure: Biannual ultrasonography — Biannual ultrasonography for HCC surveillance, performed by board-certified radiologists.
Procedure: Annual noncontrast liver MRI — Annual noncontrast liver MRI consisted of T2WI, precontrast T1WI, dual-echo image, DWI (single shot, multishot) and T2 map.
  DWI using multishot and T2 map are not included for initial MR reading.
Procedure: Contrast enhanced liver CT — In patients without report of HCC during surveillance period, contrast CT is performed 6 months after the last MR scan.

SUMMARY:
The purpose of this study is to investigate clinical feasibility of annual non-contrast magnetic resonance imaging for surveillance of hepatocellular carcinoma in high-risk group, in comparison with biannual ultrasonography.

DETAILED DESCRIPTION:
The purpose of this study is to investigate clinical feasibility of annual non-contrast magnetic resonance imaging for surveillance of hepatocellular carcinoma in high-risk group, in comparison with biannual ultrasonography. In addition, the relationship between non-contrast MR parameters and clinical manifestation of liver function is investigated.

ELIGIBILITY:
Inclusion Criteria:

* equal to or older than 40 years
* under surveillance using biannual ultrasonography (USG) and presence of liver USG within 6 months (+/- 1month)
* risk index is equal to or higher than 2.33 (Risk Index = 1.65 (if the prothrombin activity is <=75%) + 1.41 (if the age is 50 years or older) + 0.92 (if the platelet count is <=100x10(3)/mm3) + 0.74 (if the presence of HCV or HBsAg is positive)).
* signed informed consent

Exclusion Criteria:

* under 40 years
* history of HCC
* patients with pregnancy or nursing
* any contraindication of MRI
* any contraindication of CT

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
sensitivity for detecting HCC | 6 months after last patient's MRI

SECONDARY OUTCOMES:
specificity for detecting HCC | 6 months after last patient's MRI

OTHER OUTCOMES:
Apparent diffusion coefficient (ADC) | 1 month after each MR scan
  calculated value from diffusion weighted image with different protocols (conventional, simultaneous multishot)
T2 relaxation time | 1 month after MR scan
  calculated value from T2 map

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No